CLINICAL TRIAL: NCT02858817
Title: Safety and Protective Efficacy of Intravenous Immunization With Cryopreserved Plasmodium Falciparum Sporozoites Under Atovaquone/Proguanil Chemoprophylaxis
Brief Title: Safety and Protective Efficacy of IV Immunization With Cryopreserved PfSPZ Under A/P Chemoprophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Sanaria Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MALACHITE
Record Dates: First submitted 2016-07-28; First posted 2016-08-08 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2018-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Atovaquone; Proguanil; atovaquone, proguanil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 51,200 PfSPZ (Experimental): Three injections of 51,200 PfSPZ Challenge (P. falciparum strain: NF54) under chemoprophylaxis with atovaquone/proguanil 250mg/100mg (A/P) at 4 week intervals
  Interventions: Drug: atovaquone/proguanil 250mg/100mg (A/P); Biological: PfSPZ Challenge (NF54)
- 150,000 PfSPZ (Experimental): Three injections of 150,000 PfSPZ Challenge (P. falciparum strain: NF54) under chemoprophylaxis with atovaquone/proguanil 250mg/100mg (A/P) at 4 week intervals
  Interventions: Drug: atovaquone/proguanil 250mg/100mg (A/P); Biological: PfSPZ Challenge (NF54)
- Placebo (Placebo Comparator): Three injections of NaCl 0,9% solution under chemoprophylaxis with atovaquone/proguanil 250mg/100mg (A/P) at 4 week intervals
  Interventions: Drug: atovaquone/proguanil 250mg/100mg (A/P); Other: NaCl 0,9%

INTERVENTIONS:
Drug: atovaquone/proguanil 250mg/100mg (A/P) — Combination drug for chemo-prophylaxis or treatment of malaria
  Other Names: Malarone
Biological: PfSPZ Challenge (NF54) — cryo-preserved Plasmodium falciparum sporozoites injected by venous inoculation
  Arms: 150,000 PfSPZ; 51,200 PfSPZ
Other: NaCl 0,9% — 0.9% NaCl solution for injection
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Single center, randomized, placebo-controlled, double-blinded trial using PfSPZ Challenge (NF54) under A/P chemoprophylaxis for immunization and PfSPZ Challenge (NF54) and PfSPZ Challenge (7G8) for repeat CHMI.

A total of 30 adult, healthy, malaria naïve volunteers will receive three injections by Direct Venous Inoculation (DVI) of either placebo (n = 10), 51,200 PfSPZ Challenge (NF54) (n = 10), or 150,000 PfSPZ Challenge (NF54) (n = 10) under chemoprophylaxis with A/P at 4 week intervals. The placebo will be normal saline (0.9% NaCl).

Ten weeks after the last dose of PfSPZ Challenge (NF54) for immunization, volunteers will undergo first CHMI and followed until asexual blood stage parasitemia, detected by quantitative real time PCR (qPCR) or thick blood smear microscopy. If parasitemic, they will be treated with A/P (used in this case as a standard treatment regimen). In the event of no parasitemia, volunteers will be followed until Day 28 post-CHMI and will not receive A/P.

Sixteen to forty-four weeks after the last immunization, a second CHMI will be administered to assess longevity and cross-strain protection. All volunteers will be followed up to 28 days post-inoculation. Those developing parasitemia will be treated with A/P.

Volunteers of Group A will have CHMI with PfSPZ Challenge (NF54) followed by PfSPZ Challenge (7G8). Volunteers of Group B will have CHMI with PfSPZ Challenge (NF54) or PfSPZ Challenge (7G8) followed by PfSPZ Challenge (7G8). In the case that protective efficacy in Group A is ≥75% CHMI sequence will be 7G8-7G8. In the case that protective efficacy against homologous Challenge in Group A is <75%, volunteers will receive the same sequence as in Group A (NF54-7G8).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner if required.
* Residence in Tübingen or surroundings for the period of the trial.
* Women only: Must agree to practice continuous effective contraception for the duration of the study (a method which results in a low failure rate; i.e. less than 1% per year).
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local and national blood banking eligibility criteria (currently four years in Germany).
* Provision of written informed consent to receive PfSPZ Challenge for immunization and subsequently for CHMI.
* Reachable (24/7) by mobile phone during the immunization and CHMI period.
* Willingness to take A/P during immunization and a curative antimalarial regimen following CHMI.
* Agreement to stay overnight for observation during the period of intensive follow-up post-challenge if required.
* Answer all questions on the informed consent quiz correctly.
* A body mass index 18-35.

Exclusion Criteria:

* History of P.falciparum malaria.
* Planned travel to malaria endemic areas during the study period.
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrollment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin,erythromycin, fluoroquinolones, or azithromycin).
* Receipt of an investigational product in the 90 days preceding enrollment, or planned receipt during the study period.
* HIV infection.
* Any confirmed or suspected immunosuppressive or immunodeficient state (e.g. repeated and/or unusual infections),history of infection caused by opportunistic organisms any infection or combination of infections that suggest underlying immunodeficiency, history of meningitis, encephalitis, septic shock, life-threatening soft tissue infection, more than one pneumonia, asplenia and/or chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* Known (or signs consistent with) sickle cell anemia, sickle cell trait, thalassemia or thalassemia trait, glucose-6-phosphate dehydrogenase deficiency.
* Pregnancy, lactation or intention to become pregnant during the study.
* Contraindications to the use of the following antimalarial medications: A/P, artemether-lumefantrine
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60 g (men) or 40 g (women) per day or a carbohydrate deficient transferrin (CDT) level ≥2.5%.
* Suspected or known injected drug abuse in the 5 years preceding enrollment.
* Positive for hepatitis B surface antigen (HBs-antigen).
* Seropositive for hepatitis C virus (antibodies to HCV).
* Falling in moderate risk or higher categories for fatal or non-fatal cardiovascular event within 5 years (>10%) determined by non-invasive criteria for cardiac risk 84.
* Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, clinically significant arrythmias, left bundle branch block, secondary or tertiary AV block
* A QT/QTcB interval >450 ms.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* CrCL <30ml/min
* History of seizure (except uncomplicated febrile convulsion at childhood)
* Immunization with more than 3 other vaccines within the past month
* Any other significant disease, disorder, finding at medical history, biochemistry, hematology tests, urine analysis results or at clinical examination which, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Number or occurrence of related Grade 3 and 4 adverse events (AEs) and serious adverse events (SAEs) | from time of first administration of A/P until the last follow up visit, 414 days after first administration

SECONDARY OUTCOMES:
Occurrence of any related AE | from time of first administration of A/P until the last follow up visit, 414 days after first administration
Proportion of protected volunteers | From time of PfSPZ challenge administration until 28 days after PfSPZ challenge
  . Protection is defined as the absence of parasites in the peripheral blood for 28 days following first and second CHMI with PfSPZ Challenge (NF54) and PfSPZ Challenge (7G8) in volunteers receiving PfSPZ-CVac with A/P. Parasitemia is defined as at least one qPCR result above 100 parasites per mL among three positive results at least 12 hours apart or as a positive thick blood smear. Statistical testing is hierarchical: 1) protection against first CHMI, 2) protection against second CHMI.

OTHER OUTCOMES:
Time-to-parasitemia in volunteers who receive immunization using PfSPZ Challenge or placebo under A/P chemoprophylaxis and become parasitemic within 28 days following CHMI with PfSPZ Challenge (NF54) or PfSPZ Challenge (7G8). | Until 28 days after challenge
Time-to-parasitemia in placebo recipients following 2nd versus 1st CHMI (carry-over effect). | Until 28 days after challenge

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Kremsner, Prof, Principal Investigator — University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided